CLINICAL TRIAL: NCT01827904
Title: A Pivotal Study to Evaluate the Effectiveness and Safety of ExAblate Transcranial MRgFUS Thalamotomy Treatment of Medication Refractory Essential Tremor Subjects
Brief Title: ExAblate Transcranial MR Guided Focused Ultrasound for the Treatment of Essential Tremors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InSightec (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ET002
Record Dates: First submitted 2013-03-27; First posted 2013-04-10 (Estimated); Results first posted 2024-03-13 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-03

CONDITIONS: Essential Tremor
Keywords: ExAblate Transcranial MRgFUS
MeSH Terms: conditions — Essential Tremor

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Transcranial ExAblate (Experimental): Transcranial ExAblate
  Interventions: Device: Transcranial ExAblate
- Sham Transcranial ExAblate (Sham Comparator): Sham Treatment with Transcranial ExAblate
  Interventions: Device: Sham Transcranial ExAblate

INTERVENTIONS:
Device: Transcranial ExAblate
  Other Names: ExAblate; TcMRgFUS; Thalamotomy
  Arms: Transcranial ExAblate
Device: Sham Transcranial ExAblate
  Arms: Sham Transcranial ExAblate

SUMMARY:
The objective of this prospective, randomized, double-blind (to subjects, local site's blinded assessor and Tremor Core Lab assessors), crossover, multi-site, two-arm study (ExAblate treated arm Vs ExAblate Sham treated control arm) is to test the efficacy of treatment using the ExAblate Transcranial System and to further demonstrate safety in medication-refractory tremor in subjects with essential tremor (ET).

DETAILED DESCRIPTION:
This study is evaluating a new technique for performing Thalamotomy for tremor control. While current techniques have possible invasive or radiation effects, the use of ExAblate if totally non-invasive and without any radiation. After informed consent and screening, eligible subjects will be randomized to either an ExAblate treatment or an ExAblate Sham or "fake" procedure. The chance of randomization to Sham is one out of four. Subjects who are randomized to Sham Control will undergo the same procedure and follow-up visits through their Month 3 visit. After the Month 3 assessments are complete, all subjects will be unblinded and those in the Sham treated group will have the option for an actual ExAblate treatment in an unblinded fashion, as long as they still qualify for ExAblate treatment. All subjects will be followed at 6 and 12 months and for up to 5 years as directed by their doctor.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, age 22 years and older
* Subjects who are able and willing to give informed consent and able to attend all study visits
* Subjects with a diagnosis of Essential Tremor as confirmed from clinical history and examination by a neurologist or neurosurgeon specialized in movement disorder
* Subject exhibits a significant disability from their ET despite medical treatment
* Subjects should be on a stable dose of all ET medications for 30 days prior to study entry
* Subject is able to communicate sensations during the ExAblate Transcranial procedure

Exclusion Criteria:

* Subjects with unstable cardiac status
* Severe hypertension
* Subjects with standard contraindications for MR imaging such as non-MRI compatible implanted metallic devices including cardiac pacemakers, size limitations, etc.
* Known intolerance or allergies to the MRI contrast agent including advanced kidney disease or severely impaired renal function
* Significant claustrophobia that cannot be managed with mild medication
* Current medical condition resulting in abnormal bleeding and/or coagulopathy
* Receiving anticoagulant (e.g. warfarin) or antiplatelet (e.g. aspirin) therapy within one week of focused ultrasound procedure or drugs known to increase risk or hemorrhage
* History of intracranial hemorrhage
* History of multiple strokes, or a stroke within past 6 months
* Subjects who are not able or willing to tolerate the required prolonged stationary supine position during treatment
* Are participating or have participated in another clinical trial in the last 30 days
* Subjects unable to communicate with the investigator and staff
* Subjects with a history of seizures within the past year
* Subjects with brain tumors

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2021-02-24 (Actual); Study Completion 2021-02-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (5):
  - Stanford University Medical Center, Stanford, California
  - University of Maryland Medical System, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Virginia, Charlottesville, Virginia
  - Swedish Medical Center, Seattle, Washington
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada
- Tokyo Women's Medical University (TWMU), Tokyo, Japan
- Yonsei University Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Yamamoto K, Sarica C, Elias GJB, Boutet A, Germann J, Loh A, Joel SE, Bigioni L, Gwun D, Gramer R, Li SX, Zemmar A, Vetkas A, Algarni M, Devenyi G, Chakravarty M, Hynynen K, Scantlebury N, Schwartz ML, Lozano AM, Fasano A. Ipsilateral and axial tremor response to focused ultrasound thalamotomy for essential tremor: clinical outcomes and probabilistic mapping. J Neurol Neurosurg Psychiatry. 2022 Aug 22:jnnp-2021-328459. doi: 10.1136/jnnp-2021-328459. Online ahead of print. PMID 35995551
- [Derived] Cosgrove GR, Lipsman N, Lozano AM, Chang JW, Halpern C, Ghanouni P, Eisenberg H, Fishman P, Taira T, Schwartz ML, McDannold N, Hayes M, Ro S, Shah B, Gwinn R, Santini VE, Hynynen K, Elias WJ. Magnetic resonance imaging-guided focused ultrasound thalamotomy for essential tremor: 5-year follow-up results. J Neurosurg. 2022 Aug 5;138(4):1028-1033. doi: 10.3171/2022.6.JNS212483. Print 2023 Apr 1. PMID 35932269
- [Derived] Halpern CH, Santini V, Lipsman N, Lozano AM, Schwartz ML, Shah BB, Elias WJ, Cosgrove GR, Hayes MT, McDannold N, Aldrich C, Eisenberg HM, Gandhi D, Taira T, Gwinn R, Ro S, Witt J, Jung NY, Chang JW, Rosenberg J, Ghanouni P. Three-year follow-up of prospective trial of focused ultrasound thalamotomy for essential tremor. Neurology. 2019 Dec 10;93(24):e2284-e2293. doi: 10.1212/WNL.0000000000008561. Epub 2019 Nov 20. PMID 31748250
- [Derived] Elias WJ, Lipsman N, Ondo WG, Ghanouni P, Kim YG, Lee W, Schwartz M, Hynynen K, Lozano AM, Shah BB, Huss D, Dallapiazza RF, Gwinn R, Witt J, Ro S, Eisenberg HM, Fishman PS, Gandhi D, Halpern CH, Chuang R, Butts Pauly K, Tierney TS, Hayes MT, Cosgrove GR, Yamaguchi T, Abe K, Taira T, Chang JW. A Randomized Trial of Focused Ultrasound Thalamotomy for Essential Tremor. N Engl J Med. 2016 Aug 25;375(8):730-9. doi: 10.1056/NEJMoa1600159. PMID 27557301
- Available data/document: Clinical Study Report — https://www.accessdata.fda.gov/cdrh_docs/pdf15/p150038c.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: After completing the 3 Month visit subjects randomized to the Sham group were given the option to receive the Exablate thalamotomy as a rescue treatment and continue in the Crossover group. Nineteen subjects opted to continue in the Crossover group. Thus, 19 Sham Control and 19 Crossover are the same subjects. Two subjects randomized to the Exablate test group received suboptimal treatment, were retreated, and followed in the Crossover group through 12 Months resulting in N = 21.
Groups:
- Transcranial Exablate (MRgFUS) Only: The experimental design is a two-arm Test versus Sham Control study. The primary efficacy analysis was performed at Month-3 post treatment.
  Test arm: Transcranial Exablate subjects randomly assigned to the MR guided Focused Ultrasound (MRgFUS) test arm.
  Transcranial Exablate: Exablate thalamotomy for essential tremor.
- Sham Transcranial Exablate First, Then Optional Transcranial Exablate (MRgFUS): The experimental design was a two-arm Test versus Sham treatment.
  Sham arm: Sham Treatment with Transcranial Exablate subjects randomly assigned to the sham control arm.
  After completing the 3-Month study visit sham treatment control subjects could be offered the Exablate procedure as a "rescue" treatment and follow-up in the Crossover arm. This "crossover" was not a formal part of the experimental design in terms of hypothesis testing. It was analyzed separately as supplemental efficacy and safety data.
  Sham Transcranial Exablate: Exablate procedure with ultrasound energy set to zero.
- Crossover Transcranial Exablate After 3-Month Follow-Up: After completing the 3 Month visit subjects randomized to the Sham group were presented with the opportunity to receive the Exablate as a "rescue" treatment and continue in the study in the Crossover group. Nineteen subjects opted to continue in the Crossover ("rescue") group. Two subjects randomized to the Exablate test group received suboptimal treatment, were retreated, and followed in the Crossover group. Thus the total number of subjects in the initially in the Crossover group was 21.
Period: Main Study
Arm/Group | Transcranial Exablate (MRgFUS) Only | Sham Transcranial Exablate First, Then Optional Transcranial Exablate (MRgFUS) | Crossover Transcranial Exablate After 3-Month Follow-Up
Started | 56 | 20 | 0
Completed | 54 | 20 | 0
Not Completed | 2 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0
Period: Main Continuation / Crossover Phase
Arm/Group | Transcranial Exablate (MRgFUS) Only | Sham Transcranial Exablate First, Then Optional Transcranial Exablate (MRgFUS) | Crossover Transcranial Exablate After 3-Month Follow-Up
Started | 54 | 0 (After completing the Main study (primary efficacy analysis) phase subjects randomized to the Sham Control group could opt to either receive Exablate thalamotomy and continue in the Crossover group or exit the study. Nineteen out of 20 subjects randomized to the Sham Control received Exablate thalamotomy and continued follow up in the Crossover group. One subject randomized to the Sham Control completed study participation at the 3 Month visit and opted not to continue in the Crossover group.) | 21 (Nineteen out of 20 subjects initially randomized to the Sham Control group opted to receive the Exablate thalamotomy and continue follow up in the Crossover group. Two additional subjects that received sub-therapeutic Exablate thalamotomies in the Transcranical Exablate group were also re-treated and followed in the Crossover group. Thus, two subjects were followed in both the Exablate Only group and the Crossover group through the first year of follow up.)
Completed | 51 | 0 | 21
Not Completed | 3 | 0 | 0
Not completed — Alternative treatment | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Health reasons unrelated to study | 1 | 0 | 0
Period: Long-term Annual Follow-up
Arm/Group | Transcranial Exablate (MRgFUS) Only | Sham Transcranial Exablate First, Then Optional Transcranial Exablate (MRgFUS) | Crossover Transcranial Exablate After 3-Month Follow-Up
Started | 51 | 0 (After completing the 3 Month visit subjects randomized to the Sham Control group were presented with the opportunity to receive the Exablate treatment and continue in the study in the Crossover group. The Sham group went only through the 3 Month visit. Nineteen out of 20 Sham Controls opted for treatment in the Crossover Transcranial Exablate group, and the remaining subject opted for study completion at the 3 Month visit in the Sham Control group.) | 19 (The two subjects receiving suboptimal treatments in the Exablate group, retreated and followed in the Crossover group, were followed in the Exablate group after the 12 Month visit.)
Completed | 29 | 0 | 12
Not Completed | 22 | 0 | 7
Not completed — Withdrawal by Subject | 11 | 0 | 5
Not completed — Alternative Treatment | 4 | 0 | 1
Not completed — Unrelated Health Reason | 2 | 0 | 1
Not completed — Lost to Follow-up | 2 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0
Not completed — Suboptimal Treatment | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Sham Transcranial ExAblate: Sham Treatment with Transcranial ExAblate
  Sham Transcranial ExAblate
- Total: Total of all reporting groups
Arm/Group | Transcranial ExAblate | Sham Transcranial ExAblate | Total
Number analyzed (Participants) | 56 | 20 | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.8 (8.7) | 71.4 (7.3) | 71.0 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 5 | 24
  Male | 37 | 15 | 52
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 41 | 16 | 57
  Black | 0 | 0 | 0
  Asian | 14 | 4 | 18
  Hispanic | 0 | 0 | 0
  Other | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Canada | 12 | 4 | 16
  South Korea | 12 | 3 | 15
  United States | 32 | 13 | 45
Skull Density Ratio [Mean (Standard Deviation); unit: Ratio] | 0.6 (0.1) | 0.5 (0.1) | 0.6 (0.1)
CRST Tremor Motor Score [Mean (Standard Deviation); unit: Score on a Scale] — Baseline sum of upper extremity Tremor-Motor scores for the treated side from the Clinical Rating Scale for Tremor (CRST) Part A and Part B averaged across subjects. This measure of upper extremity tremor ranges from 0-32 with high scores being worse. The individual baseline scores were divided by the total score possible depending on handedness. Lower scores are better than higher scores.
  Score on a Scale | 20.16 (4.73) | 19.6 (4.51) | 20.01 (4.65)
Quality of Life for Essential Tremor (QUEST) Summary of Dimensions TOTAL Score [Mean (Standard Deviation); unit: Average of 5 Dimension Percent Scores] — Baseline Quality of Life for Essential Tremor (QUEST) TOTAL is the mean of five QUEST dimensions each as a percent of the total possible. The QUEST is a 30-item assessment with each item scored 0-4 (total min - max is 0 - 120). For each subject, each of the 5 QUEST dimension scores is a percentage (100%-0%) of total possible for each dimension. The QUEST summary of dimensions total is a mean of the five dimension scores. Lower QUEST scores are better than higher scores.
  Average of 5 Dimension Percent Scores | 42.5 (18.3) | 42.8 (19.5) | 42.6 (18.5)
CRST Part C Functional Disabilities Score [Mean (Standard Deviation); unit: Score on a Scale] — Baseline Clinical Rating Scale for Tremor (CRST) Part C is a measure of functional disability due to tremor. The Clinical Rating Scale for Tremor Part C consists of 8 items each scored from 0 to 4. Thus, the total score summed ranges from 0 to 32 (average, 0-4) and provides an overall assessment of activities of daily living. Low scores on the Clinical Rating Scale for Tremor (CRST) Part C are better. Low scores show improvement in functional disabilities compared to higher scores.
  Score on a Scale | 16.5 (4.64) | 16.1 (4.32) | 16.4 (4.53)

OUTCOME MEASURES:

1. Primary Outcome: Tremor Motor Score - Clinical Rating Scale for Tremor (CRST Part A (Upper Extremity) + Part B) Percent Change From Baseline
Description: The percent change from baseline to Month 3 follow-up in upper extremity Tremor-Motor scores for the treated side is a sub-scale of Clinical Rating Scale for Tremor (CRST) Part A and Part B sum that was used to measure treated-side upper extremity tremor changes over time. Tremor-motor scores range from 0-32 points. Individual subject's scores at Baseline and 3 Months were used to calculate percent change from baseline and averaged across subjects. High percent change from baseline is better (shows improvement).
Time Frame: Baseline, 3 Months post-treatment
Measure: Mean (95% Confidence Interval); unit: Percent Change from Baseline
Arm/Group | Transcranial ExAblate | Sham Transcranial ExAblate
Number analyzed (Participants) | 56 | 20
Percent Change from Baseline | 46.9 [40.3 to 53.5] | -0.1 [-9.6 to 9.5]
Statistical Analysis 1: Comparison: Transcranial ExAblate vs Sham Transcranial ExAblate; Note that the "Crossover" group was a rescue treatment group and not integral to the experimental design statistical analysis; Test type: Superiority — Percent change from Baseline at the 3 Month visit in the Exablate test vs. Sham control arms was tested using the t-test; p < 0.001, t-test, 1 sided; alpha = 0.05 for the hypothesis test. H0: M3ExAblate ≤ M3Sham H1: M3ExAblate > M3Sham

2. Primary Outcome: Number of Device and Procedure Related Adverse Events
Description: The cumulative sum of adverse events was followed through Year 5 of the study.
Time Frame: 5 Years post treatment.
Population: Adverse Events and Serious Adverse Events are reported in the Adverse Events Section. Nineteen of the 21 subjects were Sham group subjects opting for treatment in the Crossover group. Two out of the 21 received subtherapeutic treatment in the Transcranial Exablate group and were retreated and followed in the Crossover group.
Measure: Number; unit: Number of adverse events
Groups:
- Crossover Transcranial Exablate: After completing the 3 Month visit subjects randomized to the Sham group were presented with the opportunity to receive the Exablate treatment and continue in the study in the Crossover group. Nineteen subjects opted to continue in the Crossover group. Two subjects randomized to the Exablate test group received suboptimal treatment, were retreated, and followed in the Crossover group. Thus the total number of subjects in the initially in the Crossover group was 21.
Arm/Group | Transcranial ExAblate | Sham Transcranial ExAblate | Crossover Transcranial Exablate
Number analyzed (Participants) | 56 | 20 | 21
Number of adverse events | 184 | 26 | 75

3. Secondary Outcome: Tremor Motor Score - Clinical Rating Scale for Tremor (CRST) Part A (Upper Extremity) + Part B Percent Change From Baseline
Description: The percent change from baseline to Month 3 follow-up in upper extremity Tremor-Motor scores for the treated side is a sub-scale of Clinical Rating Scale for Tremor (CRST) Part A and Part B sum that was used to measure treated-side upper extremity tremor changes over time. Tremor-motor scores range from 0-32 points. Individual subject's scores at Baseline and Follow Up were used to calculate percent change from baseline and averaged across subjects. High percent change from baseline is better (shows improvement).
Time Frame: Baseline, 3 Months, 6 Months, 12 Months, 2, 3, 4, 5 Years post treatment
Population: Subjects randomized to the Sham control group exited the study after completing the 3 month visit. They were given the opportunity to receive the Exablate treatment and complete the follow-up visit schedule. Nineteen Sham subjects opted to continue in the Crossover. Two subjects randomized to the Exablate group received suboptimal treatment, were retreated, and continued in the Crossover.
Measure: Mean (95% Confidence Interval); unit: Percent Change from Baseline
Arm/Group | Transcranial ExAblate | Sham Transcranial ExAblate | Crossover Transcranial Exablate
Number analyzed (Participants) | 56 | 20 | 21
Percent Change from Baseline
  3 Months | 46.9 [40.3 to 53.5] | -0.1 [-9.6 to 9.5] | 53.1 [43.4 to 62.8]
  6 Months: number analyzed (Participants) | 56 | 0 | 21
  6 Months | 43.1 [36.4 to 49.9] |  | 50.7 [41.8 to 59.6]
  12 Months: number analyzed (Participants) | 56 | 0 | 16
  12 Months | 39.6 [34.0 to 45.3] |  | 47.0 [30.6 to 63.3]
  2 Years: number analyzed (Participants) | 41 | 0 | 16
  2 Years | 55.9 [48.9 to 63.0] |  | 56.2 [40.5 to 71.8]
  3 Years: number analyzed (Participants) | 38 | 0 | 15
  3 Years | 52.6 [45.5 to 59.6] |  | 53.5 [39.3 to 67.7]
  4 Years: number analyzed (Participants) | 36 | 0 | 14
  4 Years | 46.8 [37.7 to 55.8] |  | 55.5 [41.7 to 56.7]
  5 Years: number analyzed (Participants) | 29 | 0 | 12
  5 Years | 37.5 [26.3 to 48.8] |  | 50.2 [32.5 to 67.9]

4. Secondary Outcome: Clinical Rating Scale (CRST) Part A - Posture Score, Percent Change From Baseline (Pre-treatment)
Description: The Posture Score is a sub-Score of the Clinical Rating Scale for Tremor CRST Part A - Posture (Treated Side Upper Extremity Posture Score). The scores range 0-12 and higher scores indicate worse outcomes. For percent improvement compared to Baseline (pre-treatment visit) higher percents mean better outcomes.
Time Frame: Baseline, 3 Months, 6 Months, 12 Months, 2, 3, 4, 5 Years post treatment
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: Percent Change from Baseline
Arm/Group | Transcranial ExAblate | Sham Transcranial ExAblate | Crossover Transcranial Exablate
Number analyzed (Participants) | 56 | 20 | 21
Percent Change from Baseline
  3 Month: number analyzed (Participants) | 56 | 17 | 21
  3 Month | 64.3 [52.1 to 76.5] | -4.4 [-27.0 to 18.2] | 56.4 [36.6 to 76.1]
  6 Month: number analyzed (Participants) | 56 | 0 | 21
  6 Month | 62.5 [50.8 to 74.2] |  | 56.8 [36.3 to 77.2]
  12 Month: number analyzed (Participants) | 56 | 0 | 16
  12 Month | 65.5 [54.7 to 76.3] |  | 46.4 [22.3 to 70.4]
  2 Year: number analyzed (Participants) | 41 | 0 | 16
  2 Year | 73.8 [65.2 to 82.4] |  | 78.7 [68.5 to 88.8]
  3 Year: number analyzed (Participants) | 38 | 0 | 15
  3 Year | 76.8 [67.5 to 86.0] |  | 76.1 [61.6 to 90.6]
  4 Year: number analyzed (Participants) | 36 | 0 | 14
  4 Year | 72.0 [59.8 to 84.2] |  | 71.4 [56.4 to 86.4]
  5 Year: number analyzed (Participants) | 29 | 0 | 12
  5 Year | 72.0 [60.49 to 85.5] |  | 75.7 [57.8 to 93.6]

5. Secondary Outcome: Functional Disabilities - Clinical Rating Scale (CRST) for Tremor Part C Score Percent Change From Baseline
Description: 1. Subject daily functionalities: as measured by CRST Part-C (subscales) as percent change from Baseline. CRST Part-C is an 8-item score range 0-32. Higher percent change from Baseline means better outcomes.
Time Frame: Baseline, 3 Months, 6 Months, 12 Months, 2, 3, 4, 5 Years post treatment
Population: Subjects randomized to the Sham control group exited the study after completing the 3 month visit. They were given the opportunity to receive the Exablate treatment and complete the follow-up visit schedule. Nineteen Sham subjects opted to continue in the Crossover. Two subjects randomized to the Exablate group received suboptimal treatment, were retreated and continued in the Crossover.
Measure: Mean (95% Confidence Interval); unit: Percent Change from Baseline
Arm/Group | Transcranial ExAblate | Sham Transcranial ExAblate | Crossover Transcranial Exablate
Number analyzed (Participants) | 56 | 20 | 21
Percent Change from Baseline
  3 Months | 63.8 [55.3 to 72.4] | 1.8 [-6.7 to 11.1] | 74.6 [66.2 to 82.9]
  6 Months: number analyzed (Participants) | 56 | 0 | 21
  6 Months | 61.8 [53.2 to 70.4] |  | 72.1 [62.4 to 81.8]
  12 Months: number analyzed (Participants) | 56 | 0 | 18
  12 Months | 64.0 [55.2 to 72.7] |  | 68.9 [55.0 to 82.9]
  2 Years: number analyzed (Participants) | 41 | 0 | 16
  2 Years | 62.1 [53.6 to 70.6] |  | 61.9 [47.4 to 76.3]
  3 Years: number analyzed (Participants) | 38 | 0 | 15
  3 Years | 58.7 [50.1 to 67.3] |  | 51.0 [31.5 to 70.6]
  4 Years: number analyzed (Participants) | 36 | 0 | 14
  4 Years | 47.8 [35.1 to 59.9] |  | 49.5 [27.6 to 71.4]
  5 Years: number analyzed (Participants) | 29 | 0 | 12
  5 Years | 43.4 [30.8 to 56.0] |  | 51.4 [28.7 to 74.0]

6. Secondary Outcome: Quality of Life in Essential Tremor Questionnaire (QUEST) Summary Total Percent Change From Baseline
Description: The percent change from baseline to follow-up QUEST Summary Total was used to assess quality of life changes over time in tremor patients. The QUEST consists of five dimensions for each subject converted to a percent of the total (0-100%). The summary total is the average of the five dimensions. High percent change from baseline is better (shows improvement).
Time Frame: Baseline, 3 Months, 6 Months, 12 Months, 2, 3, 4, 5 Years post treatment
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: Percent Change from Baseline
Arm/Group | Transcranial ExAblate | Sham Transcranial ExAblate | Crossover Transcranial Exablate
Number analyzed (Participants) | 56 | 20 | 21
Percent Change from Baseline
  3 Months: number analyzed (Participants) | 56 | 19 | 19
  3 Months | 43.2 [34.3 to 56.3] | 5.0 [-14.9 to 36.2] | 59.2 [43.8 to 74.7]
  6 Months: number analyzed (Participants) | 56 | 0 | 20
  6 Months | 41.1 [28.8 to 53.4] |  | 58.4 [42.5 to 74.3]
  12 Months: number analyzed (Participants) | 56 | 0 | 20
  12 Months | 47.1 [34.8 to 59.5] |  | 61.5 [46.0 to 77.1]
  2 Years: number analyzed (Participants) | 41 | 0 | 16
  2 Years | 48.5 [37.4 to 59.7] |  | 49.2 [31.0 to 59.7]
  3 Years: number analyzed (Participants) | 38 | 0 | 15
  3 Years | 41.0 [25.6 to 56.3] |  | 24.3 [-19.1 to 67.6]
  4 Years: number analyzed (Participants) | 36 | 0 | 14
  4 Years | 36.9 [24.9 to 48.8] |  | 21.7 [-24.9 to 68.3]
  5 Years: number analyzed (Participants) | 29 | 0 | 12
  5 Years | 31.2 [17.9 to 44.6] |  | 16.6 [-34.2 to 67.3]

ADVERSE EVENTS:
Time Frame: Intraoperative through 5 Years. Adverse events were assessed at 3 months, 6 months, 12 months and annually for years 2 through 5.
Description: For the Exablate and Crossover Groups Adverse Events were assessed at each follow-up study visit through the 5 Year post treatment follow-up. For the Sham Group Adverse were assessed and reported through the 3 Months post treatment follow-up.
Arm/Group | Transcranial ExAblate | Sham Transcranial ExAblate | Crossover Transcranial Exablate
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/20 | 0/21
Serious Adverse Events (participants affected / at risk) | 6/56 | 0/20 | 0/21
Other Adverse Events (participants affected / at risk) | 49/56 | 6/20 | 19/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transcranial ExAblate (N=56) | Sham Transcranial ExAblate (N=20) | Crossover Transcranial Exablate (N=21)
Embolic Stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Numbness and Tingling (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Syncopal episode (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Breast cancer (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
TIA (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transcranial ExAblate (N=56) | Sham Transcranial ExAblate (N=20) | Crossover Transcranial Exablate (N=21)
Bradycardia (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Hypertentsion (Vascular disorders) | 5 (5) | 1 (1) | 2 (2)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
TIA (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 3 (3) | 0 (0) | 0 (0)
Preventricular contractions (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Sick sinus syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Vision problems (Eye disorders) | 1 (2) | 0 (0) | 0 (0)
Watering eyes (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dysgeusia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea/Vomiting (Gastrointestinal disorders) | 13 (13) | 2 (2) | 4 (4)
Increased salivation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0) | 2 (2)
Weakness (General disorders) | 1 (1) | 1 (1) | 2 (2)
Impatience (General disorders) | 1 (1) | 0 (0) | 0 (0)
Restlessness (General disorders) | 1 (1) | 0 (0) | 0 (0)
Common cold (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Flu (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Dysergia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Dysmetria (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Gait disturbance (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 0 (0)
Imbalance (Musculoskeletal and connective tissue disorders) | 10 (10) | 1 (1) | 3 (3)
Musculoskeletal weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Positional pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1) | 0 (0)
Unsteady (Musculoskeletal and connective tissue disorders) | 6 (6) | 0 (0) | 2 (2)
Anxiety (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0)
Ataxia (Nervous system disorders) | 7 (7) | 0 (0) | 4 (4)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3)
Dysesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 2 (3) | 0 (0) | 0 (0)
Dysgnosia (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Dysmetria (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Dysmnesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Grogginess (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hand tremor (untreated side) (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Involuntary movements-UE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Memory deterioration (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Numbness/Tingling (Nervous system disorders) | 18 (27) | 3 (3) | 7 (10)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2)
Slow movements (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Slurred speech (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Ankle pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Foot pain (General disorders) | 1 (1) | 1 (1) | 0 (0)
Headache (General disorders) | 14 (15) | 5 (5) | 8 (8)
Sonication-related head pain (General disorders) | 14 (14) | 0 (0) | 6 (6)
Ptosis (Product Issues) | 2 (2) | 0 (0) | 1 (1) — Stereotactic frame / Pin site related
Facial edema (Product Issues) | 1 (1) | 0 (0) | 0 (0) — Stereotactic frame / pin site related
Numbness / Tingling (Product Issues) | 1 (1) | 2 (2) | 0 (0) — Stereotactic frame / pin site related
Pin site bleeding (Product Issues) | 0 (0) | 1 (1) | 1 (1) — Stereotactic frame related
Pin site edema (Product Issues) | 1 (1) | 2 (2) | 1 (1) — Stereotactic frame related
Pin site pain (Product Issues) | 8 (8) | 3 (4) | 4 (4) — Stereotactic frame related
Pin site abrasion (Product Issues) | 2 (2) | 0 (0) | 0 (0) — Stereotactic frame related
Bruising (Product Issues) | 2 (2) | 0 (0) | 0 (0) — Stereotactic frame related
Catheter irritation (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary urgency (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
BPH (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 1 (1)
Dizziness (Ear and labyrinth disorders) | 10 (11) | 0 (0) | 3 (3)
Paroxysmal vertigo issues (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Hiccups (General disorders) | 1 (1) | 0 (0) | 0 (0)
Skin rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-08-13): https://cdn.clinicaltrials.gov/large-docs/04/NCT01827904/Prot_000.pdf
  • Statistical Analysis Plan (2014-02-10): https://cdn.clinicaltrials.gov/large-docs/04/NCT01827904/SAP_001.pdf